CLINICAL TRIAL: NCT01379781
Title: Behavioral Change in the Mother-Infant Dyad: Preventing Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Catherine Monk, Professor of Medical Psychology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #6285
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Postpartum Depression
Keywords: prevention; postpartum depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Behavior Therapy; Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Intervention for PPD (Experimental): Behavioral Intervention for PPD delivered over 3 in-person sessions.
  Interventions: Behavioral: Behavioral Intervention for PPD
- Treatment As Usual (No Intervention): Referred to Treatment in the Community.

INTERVENTIONS:
Behavioral: Behavioral Intervention for PPD — We will select a sample of pregnant women at risk for PPD, teach parenting skills to increase infant nocturnal sleep and reduce fuss/cry behavior to half of the sample during 3 perinatal visits.
  Other Names: Preventative Behavioral Intervention for PPD.
  Arms: Behavioral Intervention for PPD

SUMMARY:
Postpartum depression (PPD) is undertreated and the consequences of this are substantial for women and children. Studies show that infant cry/fuss and sleep behavior are associated with PPD, and that parenting interventions can change infant behavior, yet these findings have never been applied to PPD. In this study, the investigators are teaching parenting skills to increase infant nocturnal sleep and reduce fuss/cry behavior to women likely to develop PPD to see if the investigators can prevent the onset of this disorder.

DETAILED DESCRIPTION:
Of the over 4 million live births each year in the United States, nearly 800,000 - or 20% - of the mothers will develop major or minor depression within the first 3 months postpartum. This number dwarfs prevalence rates for gestational diabetes (2-5%) and preterm birth (12.7%). Existing clinical approaches to postpartum depression (PPD) use standard pharmacologic and psychological interventions to reduce women's symptoms. Nevertheless, PPD is undertreated, in part because women are reluctant to seek treatment due to stigma associated with mental health care and disinclination to take psychotropic medications when breastfeeding. The consequences of this are substantial. Untreated PPD is associated with diminished quality of life and significant emotional suffering for women, and, through compromised caregiving, poor outcomes in children's cognitive and social-emotional development. Although maternal risk factors for PPD are well known, protocols for prevention based on commonly used depression interventions are only beginning to be evaluated. Building on developmental data showing the profound bi-directionality of emotional and behavioral influences between mother and infant, the investigators are testing a novel PPD intervention protocol that challenges the standard, individually-focused treatment paradigm. Our intervention is based on the conceptualization of PPD as a potential disorder of the dyad, and one that can be approached through behavioral change in and affective engagement with mother and child. Studies show that infant cry/fuss and sleep behavior are associated with PPD, and that parenting interventions can change infant behavior, yet these findings have never been applied to PPD. The investigators aim to collect data on a novel PPD risk-reducing protocol based on a dyadic behavioral approach to PPD in which the investigators treat at-risk women by promoting maternally-mediated behavioral changes in their infants. The investigators will select a sample of pregnant women at risk for PPD, teach parenting skills to increase infant nocturnal sleep and reduce fuss/cry behavior to half of the sample during 3 perinatal visits, then evaluate infant behavior at 6 and 14 weeks, and maternal mood at 6, 10, and 14 weeks postpartum. The investigators will fully exploit the investigative opportunities of this intervention study by using state-of-the-art EEG and fetal monitoring to characterize early biomarkers associated with infant behavior and behavior change. This study has the potential to have a major impact on clinical research, and to transform the standard care of PPD in that (1) the intervention will have high rates of treatment compliance because (a) the protocol sessions can be incorporated into usual perinatal medical visits, (b) parenting skills will appeal to women as a non-psychiatric intervention, (c) the clinical approach will have face validity given the dyadic focus of the perinatal period; (2) its aim is prevention; (3) it fosters both maternal and child well being; (4) it will expand the risk factors for PPD to include neurobehavioral markers in the perinate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking pregnant women
* Ages 18-35
* Score of 28 or higher on the Predictive Index of Postnatal Depression
* Low to normal obstetric risk
* Before 34 weeks gestation

Exclusion Criteria:

* High Risk pregnancy
* Taking medications that affect the cardiovascular system (α blockers, β blockers, corticosteroids
* Chronic-use asthma medications (e.g. beta2-adrenoceptor agonists)
* Smoking during pregnancy
* Illicit drug/alcohol use during pregnancy
* Taking any psychotropic medications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Monk, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between July 2011 and November 2013 at Columbia University Medical Center.
Pre-assignment Details: All enrolled participants were randomized.
Groups:
- Behavioral Intervention for Postpartum Depression: Behavioral Intervention for Postpartum Depression delivered over 3 in-person sessions.
  Behavioral Intervention for Postpartum Depression: We will select a sample of pregnant women at risk for Postpartum Depression, teach parenting skills to increase infant nocturnal sleep and reduce fuss/cry behavior to half of the sample during 3 perinatal visits.
- Treatment As Usual: Referred to Treatment in the Community.
  Behavioral Intervention for PPD: We will select a sample of pregnant women at risk for PPD, teach parenting skills to increase infant nocturnal sleep and reduce fuss/cry behavior to half of the sample during 3 perinatal visits.
Period: Overall Study
Arm/Group | Behavioral Intervention for Postpartum Depression | Treatment As Usual
Started | 27 | 27
Completed | 16 | 19
Not Completed | 11 | 8
Not completed — Lost to Follow-up | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Intervention for PPD | Treatment As Usual | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.87 (6.51) | 29.60 (5.67) | 30.24 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 31
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 4 | 2 | 6
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 16 | 17 | 33
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54
Hamilton Rating Scales of Depression [Mean (Standard Deviation); unit: units on a scale] — * Assessing severity of depression; clinician rated
  * 24 questions
  * 13 items are scored on a 5 point scale ranging from 0=not present to 4=severe
  * 11 items are scored from 0-2
  * A composite score is created by the sum of the scores from all items. Scores can range from 0-74
  * 0-7: normal
  * 8-13: mild depression
  * 14-18: moderate depression
  * 19-23: severe depression
    * 24: very severe depression
      * Higher summed values indicate a greater severity of depression
  units on a scale | 18.48 (12.82) | 13.83 (17.17) | 16.16 (15.00)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scales of Depression
Description: * Assessing severity of depression; clinician rated
  * 24 questions
  * 13 items are scored on a 5 point scale ranging from 0=not present to 4=severe
  * 11 items are scored from 0-2
  * A composite score is created by the sum of the scores from all items. Scores can range from 0-74
  * 0-7: normal
  * 8-13: mild depression
  * 14-18: moderate depression
  * 19-23: severe depression
    * 24: very severe depression
      * Higher summed values indicate a greater severity of depression
Time Frame: 6 weeks postpartum
Population: Those in the analysis received both baseline and 6-week assessment sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Intervention for PPD | Treatment As Usual
Number analyzed (Participants) | 22 | 23
units on a scale | 12.09 (7.31) | 17.17 (9.81)
Statistical Analysis 1: Comparison: Behavioral Intervention for PPD; Mixed effect model was used to compare Hamilton Rating Scales of Depression (HRSD) for women who received the PREPP intervention between the pre-randomization assessment and the 6 weeks postpartum session; Test type: Superiority; p = .01, Mixed Models Analysis; Slope = -6.54

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up until 4 months postpartum.
Description: Participants were screened with the Hamilton Rating Scales for Depression and the Hamilton Anxiety Scales by a trained rater.
Arm/Group | Behavioral Intervention for PPD | Treatment As Usual
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No